CLINICAL TRIAL: NCT01630811
Title: Nuedexta for Neurobehavioral Symptoms of Adults With Autism Spectrum Disorder
Brief Title: Nuedexta for the Treatment of Adults With Autism
Acronym: Nuedexta
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sutter Health (Other)
Responsible Party: Principal Investigator, Michael Chez, MD, Principal Investigator, Sutter Health
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CHKI-Nued0911
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Results first posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-11

CONDITIONS: Autism
Keywords: Adults
MeSH Terms: conditions — Autistic Disorder | interventions — dextromethorphan - quinidine combination; Dextromethorphan; Quinidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nuedexta (Experimental): Nuedexta (Dextromethorphan hydrobromide 20 mg/quinidine sulfate 10 mg), oral, once daily
  Interventions: Drug: Nuedexta
- Placebo (Placebo Comparator): Oral, once daily
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Nuedexta — Nuedexta (Dextromethorphan hydrobromide 20 mg and quinidine sulfate 10 mg) will be given once daily for 7 days. If well-tolerated, it will be given every 12 hours for the next 7 weeks.
  Other Names: Dextromethorphan hydrobromide and quinidine sulfate
  Arms: Nuedexta
Other: Placebo — Placebo will be given once daily for 7 days.
  Arms: Placebo

SUMMARY:
Primary: Demonstrate reduced frequency and intensity of maladaptive behaviors as measured by the Aberrant Behavior Checklist (ABC) Irritability subscale in subjects given Nuedexta 8 weeks over subjects given placebo.

Secondary: Demonstrate a trend towards reduced aggressive behavior as measured by Overt Aggression Scale (OAS).

DETAILED DESCRIPTION:
This is a randomized placebo-controlled crossover study. The parents, neuropsychologists, clinical research coordinator (CRC) and PI will be blinded as to whether subjects are on placebo or Nuedexta.

Nuedexta will be given once daily for 7 days. If well-tolerated, it will be given every 12 hours for the next 7 weeks. Patients may also remain on the once-daily dose if desired.

The study will last 44 weeks. This includes 20 weeks for study enrollment, 8 weeks of treatment/placebo, 4 weeks for washout, and a second 8 week-period of treatment/placebo followed by 4 weeks of washout.

Subjects will be randomized to 8 weeks of Nuedexta/placebo. After the 8 week follow-up visit, there will be a 4 week washout period. At week 12 (second baseline), the groups will crossover for another 8 weeks of Nuedexta/placebo. Study endpoints will be measured in the both groups at weeks 8, 12, and 20. A final study visit will occur at week 24.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 60 years of age
2. Have a collateral informant who can attend visit and answer questionnaires pertaining to participant behavior
3. Diagnosis of autistic spectrum disorder based on the Diagnostic and Statistical Manual, 4th edition, Text Revised (DSM-IV-TR) criteria, developmental history, and Autism Diagnostic Observation Schedule (ADOS); or confirmed diagnosis of autism during childhood through similar methods
4. Capable of giving informed consent, or have a legal guardian capable of giving consent on the subject's behalf; patient able to assent to participate
5. Mood issues and frontal lobe type perseveration issues
6. No medication changes within 30 days and no use of new medications during the course of the study except for non-related conditions approved by the investigators

Exclusion Criteria:

1. Clinically uncontrolled epilepsy
2. Cardiovascular conditions including cardiac or structural malformation heart failure, prolonged QT interval, history of torsades de pointes, or atrioventricular (AV) block
3. Known genetic disorders, fragile x, or known brain structural abnormalities, cerebral palsy, head injury, or brain tumor
4. Known allergy to either dextromethorphan or quinidine
5. Concurrent or recent use of Monoamine oxidase inhibitor (MAOI) antidepressants pt Nuedexta
6. Concurrent use of lamotrigine or felbamate or other N-Methyl-D-aspartate (NMDA) agonists or antagonists
7. Thrombocytopenia, hepatitis, bone marrow depression or lupus-like syndrome
8. Pregnancy - sexually active females of childbearing potential must be on a reliable form of contraception
9. Other clinically significant abnormality on physical, neurological, laboratory, vital signs, that could compromise the study or be detrimental to the subject

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2012-01-24 (Actual); Primary Completion 2015-12-15 (Actual); Study Completion 2015-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael G Chez, MD, Principal Investigator — Sutter Health; Carol A Parise, PhD, Study Director — Sutter Health
Locations (1):
- Sutter Pediatric Neurology, Sacramento, California, United States

REFERENCES:
- See also: Sutter Health Research — http://checksutterfirst.org/research

RESULTS

PARTICIPANT FLOW:
Groups:
- Nuedexta First Placebo Second: Participants first received Nuedexta tablet (Dextromethorphan hydrobromide 20 mg and quinidine sulfate 10 mg) given once daily for 7 days. If well-tolerated, it will be given every 12 hours for the next 7 weeks. After a washout period of 4 weeks, they then received Placebo tablet (matching Neudexta (Dextromethorphan hydrobromide 20 mg and quinidine sulfate 10 mg) given once daily for 7 days. If well-tolerated, it will be given every 12 hours for the next 7 weeks.
- Placebo First Nuedexta Second: Participants first received Placebo tablet (matching Neudexta (Dextromethorphan hydrobromide 20 mg and quinidine sulfate 10 mg) given once daily for 7 days. If well-tolerated, it will be given every 12 hours for the next 7 weeks. After a washout period of 4 weeks, they then received Nuedexta tablet (Dextromethorphan hydrobromide 20 mg and quinidine sulfate 10 mg) given once daily for 7 days. If well-tolerated, it will be given every 12 hours for the next 7 weeks.
Period: First Intervention (8 Weeks)
Arm/Group | Nuedexta First Placebo Second | Placebo First Nuedexta Second
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0
Period: Washout (4 Weeks)
Arm/Group | Nuedexta First Placebo Second | Placebo First Nuedexta Second
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0
Period: Second Intervention (8 Weeks)
Arm/Group | Nuedexta First Placebo Second | Placebo First Nuedexta Second
Started | 7 | 6
Completed | 6 | 6
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Washout (4 Weeks)
Arm/Group | Nuedexta First Placebo Second | Placebo First Nuedexta Second
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were randomized to receive either Nuedexta tablet (Dextromethorphan hydrobromide 20 mg and quinidine sulfate 10 mg) or Placebo tablet (matching Dextromethorphan hydrobromide 20 mg and quinidine sulfate 10 mg)
Arm/Group | All Study Participants
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.68 (3.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 11
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.00 (5.86)
Autism Diagnostic Observation Schedule (ADOS) [Mean (Standard Deviation); unit: units on a scale] — The Autism Diagnostic Observation Schedule (ADOS) is a semi-structured assessment of communication, social interaction, and play (or imaginative use of materials) for individuals suspected of having autism or other pervasive developmental disorders. The total score ranges from 0 to 28 with 0 representing no abnormality present. A child is suspected to have Autism if the total ADOS score is greater than 7. The mean of the total ADOS scores is listed below.
  units on a scale | 16.31 (12.04)

OUTCOME MEASURES:

1. Primary Outcome: Change in Maladaptive Behaviors
Description: Demonstrate a change in frequency and intensity of maladaptive behaviors as measured by the Aberrant Behavior Checklist (ABC) Irritability subscale in subjects given Nuedexta 8 weeks over subjects given placebo. This checklist consists of 20 questions relating to behavior and the reported total score is on a scale from 0 to 60. A lower score can be interpreted as less frequent and/or less intense presentation of the undesirable behavior. The below values are the difference in ABC scores from baseline to 8 weeks. A negative difference indicates improved behavior.
Time Frame: Baseline and 8 weeks
Population: One subject withdrew at the time of crossover.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Oral, one time daily for 7 days.
Arm/Group | Nuedexta | Placebo
Number analyzed (Participants) | 13 | 12
units on a scale | -6.62 (11.12) | -1.08 (8.46)

2. Primary Outcome: Primary Safety Endpoints
Description: Number of serious adverse events
Time Frame: Week 0 through week 25
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Placebo tablet equivalent to Nuedexta (Dextromethorphan hydrobromide 20 mg and quinidine sulfate 10 mg) will be given once daily for 7 days. If well-tolerated, it will be given every 12 hours for the next 7 weeks.
Arm/Group | Nuedexta | Placebo
Number analyzed (Participants) | 13 | 12
Participants | 0 | 0

3. Secondary Outcome: Change in Aggressive Behavior
Description: Demonstrate a trend towards reduced aggressive behavior as measured by Overt Aggression Scale (OAS). It consists of a scale from 0 - 40, and a lower score can be interpreted as less frequent and/or less intense presentation of the undesirable behavior. Reported is the mean difference in scores from baseline to 8 weeks. A positive score indicates more aggressive behavior and a negative score indicates less aggressive behavior.
Time Frame: Baseline and 8 weeks
Population: One subject withdrew at the time of crossover.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Nuedexta: Nuedexta (Dextromethorphan hydrobromide 20 mg and quinidine sulfate 10 mg) will be given once daily for 7 days. If well-tolerated, it will be given every 12 hours for the next 7 weeks.
Arm/Group | Nuedexta | Placebo
Number analyzed (Participants) | 13 | 12
units on a scale | -1.92 (2.78) | 0.08 (1.88)

ADVERSE EVENTS:
Time Frame: Eight weeks for each intervention with 4 weeks washout in between interventions and at the end (total 24 weeks).
Description: Safety population included all participants who received at least one dose of intervention.
Arm/Group | Nuedexta | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No